CLINICAL TRIAL: NCT06543498
Title: Pilot Study - The Effect of Bioactive Compounds N-trans-Caffeoyltyramine (NCT) and N-trans-Feruloyltyramine (NFT) on Intestinal Barrier Function in Participants With Irritable Bowel Syndrom With Diarrhoea
Brief Title: The Effect of Dietary Supplementation on Intestinal Barrier Function in IBS-D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr Anthony Hobson (Other)
Responsible Party: Sponsor-Investigator, Dr Anthony Hobson, Chief Investigator, The Functional Gut Clinic
Organization: The Functional Gut Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FGC-24-003
Record Dates: First submitted 2024-07-23; First posted 2024-08-09 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Irritable Bowel Syndrome With Diarrhea
MeSH Terms: interventions — Diet Records

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NCT and NFT (Active Comparator): 21 days of 1x capsule per day. Dosage 120mg.
  Interventions: Diagnostic Test: Lactulose/Mannitol Ratio Test; Diagnostic Test: Serum biomarkers of intestinal permeability; Other: Rome IV questionnaire; Other: Irritable bowel severity scoring system; Other: Bowel Habit diary; Other: 3 day dietary record; Dietary Supplement: NCT and NFT
- Placebo (Placebo Comparator): 21 days of 1x placebo capsule per day
  Interventions: Diagnostic Test: Lactulose/Mannitol Ratio Test; Diagnostic Test: Serum biomarkers of intestinal permeability; Other: Rome IV questionnaire; Other: Irritable bowel severity scoring system; Other: Bowel Habit diary; Other: 3 day dietary record; Other: Placebo

INTERVENTIONS:
Diagnostic Test: Lactulose/Mannitol Ratio Test — To test for gut permeability, Urine collected over 8hrs after ingestion of lactulose/mannitol drink.
Diagnostic Test: Serum biomarkers of intestinal permeability — Phlebotomy and subsequent lab tests to analyse concentration of LPS, LPB, sCD14, Zonulin and Occludin.
Other: Rome IV questionnaire — Diagnositic questionnaire for IBS-D
Other: Irritable bowel severity scoring system — Questionnaire to determine severity of abdominal and bowel symptoms
Other: Bowel Habit diary — Assess bowel habit at baseline and changes in bowel habit over the study
Other: 3 day dietary record — Used to verify compliance to exclusion criteria #5.
Dietary Supplement: NCT and NFT — N-transcaffeoyltyramine and N-transferuloyltyramine supplement taken once per day.
  Arms: NCT and NFT
Other: Placebo — Placebo supplement taken once per day.
  Arms: Placebo

SUMMARY:
Many people suffer from Irritable Bowel Syndrome (IBS) every year in the UK. Depending on the stool consistency, IBS can be classified as IBS with diarrhoea (IBS-D), IBS with constipation (IBS-C), or mixed IBS (IBS-M). Around 24% of those suffering with IBS have the diarrhoea variant.

IBS-D has been shown to greatly impact sufferers' quality of life and there is currently a lack of well tolerated therapies to treat this condition. Therefore, it is of upmost important to find safe and effective non-pharmacological treatments for this condition.

Two natural compounds which may interact with the body NCT and NFT have been identified in a range of edible sources and can be involved in processes that help maintain an effective gut barrier and therefore potentially help treat a leaky gut.

This research study aims to examine the effectiveness of these compounds, NCT and NFT in combination compared to a placebo (capsule that looks the same as the study product but contains no active study ingredient) capsule on gut barrier function in individuals suffering from IBS-D.

ELIGIBILITY:
Inclusion Criteria:

1. Participant has provided written informed consent before participating in the study after being given a full description of the study and prior to any study-specific procedures being performed.
2. Participant has irritable bowel syndrome with diarrhoea (IBS-D), as defined by the Rome IV criteria, confirmed by bowel diary.
3. Participant has an IBS-SSS score of >175
4. LPS at screening >0.21 ng/ml.
5. Participant is a male or non-pregnant female and is 18-70 years of age
6. If WOCBP participant is willing to adhere to one of the following methods of contraception i) Hormonal contraception e.g. the 'pill' or an implant ii) Intrauterine device (IUD) iii) Intrauterine hormone-releasing system (IUS) iv) Hysterectomy v) Vasectomised partner vi) Sexual abstinence (if it is in line with your preferred and usual lifestyle).
7. Participant can communicate well with the Investigator and to comply with the requirements for the entire study.
8. Participant has capacity to understand written English.
9. Participant has a body mass index (BMI) of 18.5 - 39.9kg/m2 (bounds included).
10. Participant agrees to follow all pre-test preparation before L/M testing.

Exclusion Criteria:

1. Prior abdominal surgery other than appendectomy, tubal ligation, hysterectomy or cholecystectomy.
2. Participated in a trial of an investigational medical product or medical device in the last 28 days.
3. Females who report to be pregnant or lactating
4. Unwilling to maintain stable doses of permitted concomitant medication.
5. Unwilling to maintain a stable diet for the duration of the trial.
6. Being in the opinion of the investigator unsuitable
7. Insufficient knowledge of English to complete the daily bowel diary and food diary.
8. Hypersensitivity to any component of the supplement
9. Hypersensitivity or known allergy to lactulose or mannitol.
10. Consumption of oral antibiotics in the last 2 weeks.
11. NSAIDs for 2 weeks prior to and during the entire 21 day study period. Participant should not be a chronic NSAID user (>1 day/week).
12. Participants who have received bowel preparation for investigative procedures in the 4 weeks prior to the study.
13. Diabetes mellitus (type 1).
14. Participants with known hepatic disease.
15. Inflammatory bowel disease (Crohn's/Colitis) or coeliac disease.
16. Gastrointestinal infection in the past 4 weeks.
17. Any other condition, deemed by the investigator, that may be causing their symptoms.
18. Participant is involved in this study as an Investigator, sub-Investigator, study coordinator, other study staff, or Sponsor member.
19. Participant is unable to adhere to withholding in endurance exercise, such as >45 minutes of high intensity running, cycling, rowing etc, from the screening phone call to the end of study visit.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-01-13 (Actual); Study Completion 2025-01-13 (Actual)

PRIMARY OUTCOMES:
Change in intestinal permeability | Day 0 vs Day 21
  Lactulose mannitol ratio change in urine from baseline to end of treatment

SECONDARY OUTCOMES:
Serum LPS | Day 0 vs Day 21
  Comparison of start to end of study between active and placebo groups
Serum LPB | Day 0 vs Day 21
  Comparison of start to end of study between active and placebo groups
Serum sCD14 | Day 0 vs Day 21
  Comparison of start to end of study between active and placebo groups
Serum Zonulin | Day 0 vs Day 21
  Comparison of start to end of study between active and placebo groups
Serum Occludin | Day 0 vs Day 21
  Comparison of start to end of study between active and placebo groups
Serum LCN12 | Day 0 vs Day 21
  Comparison of start to end of study between active and placebo groups
Rescue medication | Mean Day 0-6 vs Mean Day 15-21
  Use of rescue medication - number of days required during treatment period first week vs last week.
Loperamide utilisation | Mean Day 0-6 vs Mean Day 15-21
  Difference between active and placebo groups
Irritable bowel severity scoring system | Day 0 vs Day 21
  Change in mean score at end of treatment vs start. Minimum score 0, maximum 500. Higher score indicates worse symptoms.
Stool consistency | Day -14 to -1 vs Day 0 to 21
  Average number of days of Bristol stool scale 6-7 stools during screening vs treatment period
Stool consistency | Mean Day 0-6 vs Mean Day 15-21
  Average number of days of Bristol stool scale 6-7 stools comparison of first vs last week of treatment period
Stool frequency | Day -14 to -1 vs Day 0 to 21
  Comparison of mean number of bowel movements per day screening vs treatment period.
Stool frequency | Mean Day 0-6 vs Mean Day 15-21
  Comparison of mean number of bowel movements per day first vs last week of treatment period.
Bloating | Day -14 to -1 vs Day 0 to 21
  Comparison of mean daily bloating score screening vs treatment period. Minimum score is 0, Maximum score is 3. Higher score indicates more symptoms.
Bloating | Mean Day 0-6 vs Mean Day 15-21
  Comparison of mean daily bloating score first vs last week of treatment period. Minimum score is 0, Maximum score is 3. Higher score indicates more symptoms.
Abdominal pain | Day -14 to -1 vs Day 0 to 21
  Comparison of mean daily abdominal pain score screening vs treatment period. Minimum score is 0, Maximum score is 3. Higher score indicates more symptoms.
Abdominal pain | Mean Day 0-6 vs Mean Day 15-21
  Comparison of mean daily abdominal pain score first vs last week of treatment period. Minimum score is 0, Maximum score is 3. Higher score indicates more symptoms.

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - The Functional Gut Clinic, London
  - The Functional Gut Clinic, Manchester

IPD SHARING:
Plan to Share IPD: No